CLINICAL TRIAL: NCT00212160
Title: The Role of the Omentum in the Treatment of Morbid Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Naji Abumrad, Chairman, Department of Surgery, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: IRB #040572; R01DK070860 (NIH); 3R01DK070860-01S1 (NIH); NCT00247598 (obsolete NCT alias)
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2017-02-01 (Estimated); Status verified 2017-01

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- RYGB with omentectomy (Experimental): Subjects undergoing RYGB will be randomized to also have the greater omentum removed at the time of surgery.
  Interventions: Procedure: omentectomy
- RYGB without omentectomy (No Intervention): Subjects undergoing RYGB will be randomized to NOT have the greater omentum removed at the time of surgery.
- Normal body weight (No Intervention): Healthy normal weight subjects studied via hyperinsulinemic-euglycemic clamp to obtain reference values for insulin sensitivity and other metabolic parameters.
- Tissue samples (No Intervention): Tissue samples (omental fat, subcutaneous fat, muscle,and blood)are obtained from subjects of varying weights during abdominal surgery in order to compare various parameters, including inflammation, oxidative stress, and gene expression, among tissues across weight classes.

INTERVENTIONS:
Procedure: omentectomy — RYGB with omentectomy
  Arms: RYGB with omentectomy

SUMMARY:
The purpose of this research is to determine some of the reasons that blood sugar and insulin levels improve after bariatric surgery but before weight loss begins, as well as why people respond differently to weight loss surgery. It will also examine whether removing the fat around the stomach and large intestine (the omentum) will improve weight loss. Finally, it will see why there are differences between Whites and African Americans who have weight loss surgery.

DETAILED DESCRIPTION:
The purpose of this research is to tease out the mechanisms related to changes in insulin sensitivity, metabolism, hormones, and body composition following bariatric surgery. Because preliminary data indicate differing responses to this surgery, both Caucasian and African American adults, scheduled for RYGB, are being recruited to participate. It is believed that the omentum contributes to hepatic insulin resistance, both because of the increased delivery of NEFAs via the portal vein, and the increased production of cytokines. Because of this, it is postulated that removing the omentum as part of bariatric surgery will speed up the reversal of insulin resistance and diminish racial differences in response to the surgery.

Data are derived from tissue and blood samples obtained operatively (from individuals having bariatric surgery and other abdominal operations), as well as during hyperinsulinemic-euglycemic clamps, from indirect calorimetry, DEXA, Health-related Quality of Life surveys, and 24-hour urine samples. There were 66 participants randomized to omentectomy/no omentectomy. A post hoc data power analysis determined that this number of subjects is sufficient for data analysis.

ELIGIBILITY:
Inclusion Criteria:

* BMI > 40
* BMI > 35 with co-morbidities
* normal creatinine/liver labs
* insurance approval for RYGB or resources to self-pay
* proximity to Nashville, TN

Exclusion Criteria:

* use of anticoagulants, steroids, therapeutic niacin
* previous bariatric surgery

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2005-01 (Actual); Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
change in insulin sensitivity | 5 year

SECONDARY OUTCOMES:
Weight loss | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Naji N Abumrad, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

REFERENCES:
- [Result] Fabbrini E, Tamboli RA, Magkos F, Marks-Shulman PA, Eckhauser AW, Richards WO, Klein S, Abumrad NN. Surgical removal of omental fat does not improve insulin sensitivity and cardiovascular risk factors in obese adults. Gastroenterology. 2010 Aug;139(2):448-55. doi: 10.1053/j.gastro.2010.04.056. Epub 2010 May 7. PMID 20457158
- [Result] Saliba J, Kasim NR, Tamboli RA, Isbell JM, Marks P, Feurer ID, Ikizler A, Abumrad NN. Roux-en-Y gastric bypass reverses renal glomerular but not tubular abnormalities in excessively obese diabetics. Surgery. 2010 Feb;147(2):282-7. doi: 10.1016/j.surg.2009.09.017. Epub 2009 Dec 11. PMID 20004430
- [Result] Hajri T, Tao H, Wattacheril J, Marks-Shulman P, Abumrad NN. Regulation of adiponectin production by insulin: interactions with tumor necrosis factor-alpha and interleukin-6. Am J Physiol Endocrinol Metab. 2011 Feb;300(2):E350-60. doi: 10.1152/ajpendo.00307.2010. Epub 2010 Nov 9. PMID 21062957
- [Result] Albaugh VL, Flynn CR, Cai S, Xiao Y, Tamboli RA, Abumrad NN. Early Increases in Bile Acids Post Roux-en-Y Gastric Bypass Are Driven by Insulin-Sensitizing, Secondary Bile Acids. J Clin Endocrinol Metab. 2015 Sep;100(9):E1225-33. doi: 10.1210/jc.2015-2467. Epub 2015 Jul 21. PMID 26196952
- [Result] Knuth ND, Johannsen DL, Tamboli RA, Marks-Shulman PA, Huizenga R, Chen KY, Abumrad NN, Ravussin E, Hall KD. Metabolic adaptation following massive weight loss is related to the degree of energy imbalance and changes in circulating leptin. Obesity (Silver Spring). 2014 Dec;22(12):2563-9. doi: 10.1002/oby.20900. Epub 2014 Sep 19. PMID 25236175
- [Result] Tamboli RA, Breitman I, Marks-Shulman PA, Jabbour K, Melvin W, Williams B, Clements RH, Feurer ID, Abumrad NN. Early weight regain after gastric bypass does not affect insulin sensitivity but is associated with elevated ghrelin. Obesity (Silver Spring). 2014 Jul;22(7):1617-22. doi: 10.1002/oby.20776. Epub 2014 Apr 29. PMID 24777992
- [Result] Tamboli RA, Hajri T, Jiang A, Marks-Shulman PA, Williams DB, Clements RH, Melvin W, Bowen BP, Shyr Y, Abumrad NN, Flynn CR. Reduction in inflammatory gene expression in skeletal muscle from Roux-en-Y gastric bypass patients randomized to omentectomy. PLoS One. 2011;6(12):e28577. doi: 10.1371/journal.pone.0028577. Epub 2011 Dec 16. PMID 22194858
- [Result] Tamboli RA, Hossain HA, Marks PA, Eckhauser AW, Rathmacher JA, Phillips SE, Buchowski MS, Chen KY, Abumrad NN. Body composition and energy metabolism following Roux-en-Y gastric bypass surgery. Obesity (Silver Spring). 2010 Sep;18(9):1718-24. doi: 10.1038/oby.2010.89. Epub 2010 Apr 22. PMID 20414197
- [Derived] Dunn JP, Abumrad NN, Breitman I, Marks-Shulman PA, Flynn CR, Jabbour K, Feurer ID, Tamboli RA. Hepatic and peripheral insulin sensitivity and diabetes remission at 1 month after Roux-en-Y gastric bypass surgery in patients randomized to omentectomy. Diabetes Care. 2012 Jan;35(1):137-42. doi: 10.2337/dc11-1383. Epub 2011 Oct 31. PMID 22040841